CLINICAL TRIAL: NCT02778438
Title: REINVENT:A Validation Study of the Novel Application of Telehealth in Clinical Drug Development in Subjects With Mild Cognitive Deficits
Brief Title: A Validation Study of the Novel Application of Telehealth in Clinical Drug Development in Subjects With Mild Cognitive Deficits
Acronym: REINVENT
Status: Completed | Type: Observational
Sponsor: Quintiles, Inc. (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: REI-001
Record Dates: First submitted 2016-04-27; First posted 2016-05-19 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-05

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
REINVENT is a non-interventional, multi-center, research network-based cross-over study evaluating the potential utility of a telehealth platform in improving the efficiency of clinical trials. The study aims to enroll 30 subjects from primary care practices coordinated through a single main study site. Potential subjects will be screened and randomized (1:1) at Visit 1 into a 2-period crossover design study where 4 standard cognitive outcome measures are administered at Visits 2 (Day 30 ±7) and 3 (Day 90 ±7), either remotely or during an in-person visit.

DETAILED DESCRIPTION:
Mobile platforms have been leveraged in a variety of industries to drive dramatic efficiency gains. The technology enables redesign of key processes allowing for the more efficient use of labor and capital leading to better performance outcomes. Telehealth is the use of electronic information and mobile telecommunications technologies to support long-distance clinical health care, patient and professional health-related education, public health and health administration. Much of the focus for the Institute of Medicine and other government agencies has been the application of telehealth to improve access to healthcare and specialized expertise by extending the reach of scarce resources to underserved populations. These platforms are also routinely deployed as disease management tools. A natural extension of these aims is the use of telehealth in the clinical development process, where both improved efficiency and the ability to be more inclusive of a broader patient population are critical steps in modernizing the clinical trial.

REINVENT is a non-interventional, multi-center, research network-based cross-over study evaluating the potential utility of a telehealth platform in improving the efficiency of clinical trials. The study aims to enroll 30 subjects from between 9 and 11 qualified Radiant Clinical Research primary care physicians (PCP), coordinated through a single main study site. Potential subjects will be screened and randomized (1:1) at Visit 1 into a 2-period crossover design study where 4 standard cognitive outcome measures are administered at Visits 2 (Day 30 ±7) and 3 (Day 90 ±7), either remotely or during an in-person visit. A 60-day interval is required between Visits 2 and 3 to reduce learning effects commonly observed with repeated administration of cognitive assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age at screening 50 to 85 years, inclusive, at the time of informed consent.
* Diagnosis of mild cognitive deficits due to AD based on the core clinical diagnostic criteria of the National Institute of Aging and Alzheimer's Association (Albert 2011; McKhann 2011) and reviewed centrally by a main study site Principal Investigator
* Mini Mental State Examination (MMSE) score of 24-27, inclusive at screening
* Subject (or legally authorized representative) is willing and able to provide written informed consent
* Existence of a reliable study partner (i.e., someone who spends at least 2 days a week with the subject) or caregiver who is willing to attend study visits with the subject
* Willing and able to travel to the main study site (via provided transportation) for either Visit 2 or Visit 3

Exclusion Criteria:

* Any medical or neurological condition (other than AD) that might be a contributing cause of the subject's cognitive impairment
* Have had a stroke or transient ischemic attack (TIA) or unexplained loss of consciousness in the past 1 year
* Clinically significant psychiatric illness in past 6 months
* Relevant brain hemorrhage, bleeding disorder and cerebrovascular abnormalities
* Alcohol or substance abuse in past 1 year
* History of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class III or IV), or clinically significant conduction abnormalities (e.g., unstable atrial fibrillation) within 1 year prior to Screening.
* Uncontrolled hypertension defined as a systolic blood pressure [SBP]/diastolic blood pressure [DBP] readings > 165/100 mmHg at Screening, or persistent SBP/DBP readings prior to enrollment that in the opinion of the Investigator are indicative of chronic uncontrolled hypertension.
* Any medications that, in the opinion of the Investigator, may contribute to cognitive impairment, or impair the subject's ability to perform cognitive testing.
* Use of allowed chronic medications at doses that have not been stable for at least 4 weeks prior to Screening Visit 1 or use of AD medications (including but not limited to donepezil, rivastigmine, galantamine, tacrine, and memantine) at doses that have not been stable for at least 8 weeks prior to Screening Visit 1.
* Participation in any interventional clinical research study within 30 days prior to screening, or during study conduct
* In the opinion of the Investigator, presence of any other clinical conditions (e.g., life expectancy, co-existing disease) or other characteristics that would likely interfere with completion of the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 subjects with mild cognitive impairment due to AD, based on core clinical diagnostic criteria from the National Institute on Aging and Alzheimer's Association workgroup [Albert 2011]
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Mini Mental State Examination | 30 days, 90 days
Change in Clinical Dementia Rating Sum of Boxes | 30 days, 90 days
Change in Alzheimer's Disease Assessment Scale-Cognitive Subscale | 30 days, 90 days
Change in Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory (Mild Cognitive Impairment version) | 30 days, 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Shy, MD, Principal Investigator — Clinical Research Advantage, Inc / Neurological Physicians of Arizona, Inc
Locations (1):
- Clinical Research Advantage, Inc / Neurological Physicians of Arizona, Inc, Gilbert, Arizona, United States

IPD SHARING:
Plan to Share IPD: No